CLINICAL TRIAL: NCT00842374
Title: Single Center Registry of Non-STEMI Acute Coronary Syndrome Patients Treated With Bivalirudin
Status: Completed | Type: Observational
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: The Medicines Company (Industry)
Responsible Party: Sponsor
Other Study IDs: acs001
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Non-STEMI Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-STEMI ACS

SUMMARY:
This is a registry of patients with non ST segment elevation Myocardial Infarction (heart attack) and/or unstable acute coronary artery syndrome treated with a standardized protocol including Bivalirudin.

Data will be collected on diagnosis, treatment and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Chest pain or symptoms believed to be an anginal equivalent and representing myocardial ischemia, lasting at least 10 minutes within the past 24 hours
* Having any one of the following:

  1. Ischemic changes on ECG: ST depression >0.5 mm OR T wave inversion >2 mm
  2. Positive cardiac markers
  3. New onset CHF presumed secondary to ischemia
  4. Pulmonary edema
  5. Known coronary artery disease with typical symptoms
  6. Hemodynamic instability
  7. Sustained ventricular tachycardia

Exclusion Criteria:

* For the purpose of the SSDI, patients will be excluded if we are unable to obtain their Social Security Number.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of MACE defined as any one of the following: • Acute myocardial infarction/reinfarction • Ischemia-driven unplanned revascularizations • Stroke • All cause Mortality | 30 days

SECONDARY OUTCOMES:
Rehospitalization for ACS | 30 days
All cause mortality | 30 days, one year and up to 5 years
Major Bleeding | in hospital and at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: David M Larson, MD, Principal Investigator — Minneapolis Heart Institute Foundation
Locations (1):
- Ridgeview Medical Center, Waconia, Minnesota, United States

REFERENCES:
- [Background] Gibler WB, Cannon CP, Blomkalns AL, Char DM, Drew BJ, Hollander JE, Jaffe AS, Jesse RL, Newby LK, Ohman EM, Peterson ED, Pollack CV; American Heart Association Council on Clinical Cardiology (Subcommittee on Acute Cardiac Care); Council on Cardiovascular Nursing, and Quality of Care and Outcomes Research Interdisciplinary Working Group; Society of Chest Pain Centers. Practical implementation of the guidelines for unstable angina/non-ST-segment elevation myocardial infarction in the emergency department: a scientific statement from the American Heart Association Council on Clinical Cardiology (Subcommittee on Acute Cardiac Care), Council on Cardiovascular Nursing, and Quality of Care and Outcomes Research Interdisciplinary Working Group, in Collaboration With the Society of Chest Pain Centers. Circulation. 2005 May 24;111(20):2699-710. doi: 10.1161/01.CIR.0000165556.44271.BE. PMID 15911720
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr, Jacobs AK, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction); American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Academic Emergency Medicine. ACC/AHA 2007 guidelines for the management of patients with unstable angina/non ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction): developed in collaboration with the American College of Emergency Physicians, the Society for Cardiovascular Angiography and Interventions, and the Society of Thoracic Surgeons: endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic Emergency Medicine. Circulation. 2007 Aug 14;116(7):e148-304. doi: 10.1161/CIRCULATIONAHA.107.181940. Epub 2007 Aug 6. No abstract available. PMID 17679616
- [Background] Henry TD, Sharkey SW, Burke MN, Chavez IJ, Graham KJ, Henry CR, Lips DL, Madison JD, Menssen KM, Mooney MR, Newell MC, Pedersen WR, Poulose AK, Traverse JH, Unger BT, Wang YL, Larson DM. A regional system to provide timely access to percutaneous coronary intervention for ST-elevation myocardial infarction. Circulation. 2007 Aug 14;116(7):721-8. doi: 10.1161/CIRCULATIONAHA.107.694141. Epub 2007 Aug 1. PMID 17673457
- [Background] Henry TD, Unger BT, Sharkey SW, Lips DL, Pedersen WR, Madison JD, Mooney MR, Flygenring BP, Larson DM. Design of a standardized system for transfer of patients with ST-elevation myocardial infarction for percutaneous coronary intervention. Am Heart J. 2005 Sep;150(3):373-84. doi: 10.1016/j.ahj.2005.01.059. PMID 16169311
- [Background] Stone GW, Bertrand M, Colombo A, Dangas G, Farkouh ME, Feit F, Lansky AJ, Lincoff AM, Mehran R, Moses JW, Ohman M, White HD. Acute Catheterization and Urgent Intervention Triage strategY (ACUITY) trial: study design and rationale. Am Heart J. 2004 Nov;148(5):764-75. doi: 10.1016/j.ahj.2004.04.036. PMID 15523305
- See also: Minneapolis Heart Institute Foundation — http://www.mplsheart.org/